CLINICAL TRIAL: NCT03713034
Title: An Accessible Digital Intervention to Promote the Use of School-based Health Centers and to Empower Adolescents With Their Sexual Health
Brief Title: An Accessible Digital Intervention to Promote HIV Testing/Counseling and Prevention Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1604017531_II; 5R42HD088317-03 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: HIV Prevention
Keywords: HIV testing and counseling (HTC)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Game (Experimental): PlayTest! is an interactive world in which the player, using an avatar they have created, "travels" through life in high school. They face challenges that bring different risks and benefits, requiring them to practice decision-making skills. The player learns skills that aim to empower them to make safe choices in situations that may otherwise increase their risk for HIV/STI infection. The game also provides opportunities for the player to practice advocating for their health by modeling a conversation with a medical professional. PlayTest! incorporates evidence-based tools for behavior change including social learning theory and self-efficacy. message framing, motivational interviewing to identify the variables that must be targeted to increase HTC among adolescents.
  Interventions: Other: PlayTest!
- Control Game (Active Comparator): Some examples of control games that participants could play are: The Sims, Harry Potter, Subway Surfer, Tetris. The control games contained not relevant content related to HIV Testing and Counseling.
  Interventions: Other: Control games

INTERVENTIONS:
Other: PlayTest! — Participants in the PlayTest! intervention arm played the game on their assigned iPads once per week for an hour over the course of 4-5 weeks.
  Arms: Active Game
Other: Control games — Participants in the control arm played the games on their assigned iPads once per week for an hour over the course of 4-5 weeks.
  Arms: Control Game

SUMMARY:
This is Phase II of a study previously registered on ClinicalTrials.gov (NCT02812329). Phase II focuses on adapting and expanding the reach of a previously developed video game aimed at HIV prevention. The game will be adapted to include web access/distribution and be evaluated using a randomized controlled trial.

DETAILED DESCRIPTION:
The specific aims for Phase II of this study are to:

Further adapt and expand our culturally and socially-tailored videogame to have a greater focus on HIV testing and counseling (HTC) in addition to HIV prevention in an older age group of 14-18 year old boys and girls.

This will be accomplished by refining the conceptual model of the theoretical mechanisms of behavior change to be applied specifically within the game. New content will be created with additional input from 4 focus groups of 5 adolescents each (n = 20, aged 14-18) and these participants will also play-test the game. In addition, this model will inform new intervention manuals ("Game Playbooks") targeting these new outcomes. Building the new content from focus groups into the game are intended to adapt and expand its scope.

A system will be established for the newly adapted game for web access/distribution and program integration. Work will continue with commercialization partners on widespread distribution of the adapted game.

The final piece of the study will be to conduct a randomized controlled trial in 296 adolescents (aged 14-18) to evaluate the acceptability and efficacy of the adapted game on its new web-based platform compared with a set of control games.

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in a web-based videogame (willing to sit for 60 minutes/session to play the game)
* Have not been tested for HIV in the past year
* Ability to provide assent/parental/guardian consent+
* Have a completed and signed enrollment form for their school's health clinic allowing them, if they choose, to access the clinic for testing and health care

  * Students can be older than 18 as long as they were 18 or younger at the time of signing consent

Exclusion Criteria:

* Failure to meet any of the eligibility criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Fiellin, MD, Principal Investigator — Associate Professor of Medicine (General Medicine) and in the Child Study Center; Director, Yale Center for Health & Learning Games; Director, play2PREVENT Lab at Yale
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PlayTest! Game: Participants who were randomized to the intervention arm of the project, played the PlayTest! game on their assigned iPad, once per week for an hour, over the course of 4-5 weeks.
- Control Games: Participants who were randomized to the control arm were provided a menu of attention control games to choose from on their iPads that had no content related to HTC or HIV. Some examples of control games that participants could play are: The Sims, Harry Potter, Subway Surfer, Tetris. Participants played the choice of control games on their assigned iPad, once per week for and hour, over the course of 4-5 weeks.
Period: Overall Study
Arm/Group | PlayTest! Game | Control Games
Started | 150 | 146
Completed | 145 | 142
Not Completed | 5 | 4
Not completed — Withdrawn by staff for incomplete consent forms | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- PlayTest! Game: PlayTest! is an interactive world in which the player, using an avatar they have created, "travels" through life in high school. They face challenges that bring different risks and benefits, requiring them to practice decision-making skills. The player learns skills that aim to empower them to make safe choices in situations that may otherwise increase their risk for HIV/STI infection. The game also provides opportunities for the player to practice advocating for their health by modeling a conversation with a medical professional. PlayTest! incorporates evidence-based tools for behavior change including social learning theory and self-efficacy. message framing, motivational interviewing to identify the variables that must be targeted to increase HTC among adolescents.
  Participants who were randomized to the intervention arm of the project, played the PlayTest! game on their assigned iPad, once per week for an hour, over the course of 4-5 weeks.
- Total: Total of all reporting groups
Arm/Group | PlayTest! Game | Control Games | Total
Number analyzed (Participants) | 145 | 142 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.39 (1.24) | 15.45 (1.25) | 15.42 (1.24)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 73 | 68 | 141
  Gender: Female | 68 | 69 | 137
  Gender: Self-Described | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Native American | 4 | 4 | 8
  Asian or Pacific Islander | 8 | 5 | 13
  Black or African American | 57 | 58 | 115
  Multi-racial | 15 | 17 | 32
  Other | 27 | 23 | 50
  White | 34 | 35 | 69
Region of Enrollment [Number; unit: participants]
  United States | 145 | 142 | 287

OUTCOME MEASURES:

1. Primary Outcome: Attitudes Around HIV Testing and Counseling
Description: HTC attitudes were assessed with 7 items (e.g., "I feel it is important for me to get tested for HIV"). The items were scored on a 5-point scale ranging from - 2 (strongly disagree) to +2 (strongly agree) with positive values indicating healthier attitudes towards HTC. Participants had the option to respond "not sure" which was given a neutral score of 0. A mean of the seven items was calculated for each participant. A few items were reverse coded, because the lower value was indicating healthier attitudes. Not sure was coded as a neutral option. Higher scores equal more positive attitudes toward HIV testing and counseling.
Time Frame: Baseline, 4 weeks, 3 months and 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
score on a scale
  Baseline | 0.33 (0.65) | 0.33 (0.70)
  4 Weeks | 0.74 (0.66) | 0.26 (0.59)
  3 Months | 0.67 (0.64) | 0.24 (0.63)
  6 Months | 0.65 (0.66) | 0.27 (0.62)

2. Secondary Outcome: Intentions to Get Tested for HIV
Description: Intentions were assessed with 7 items (e.g., "I intend to get tested for HIV at some point in the next 3 months" and "I intend to use a school-based health center to get tested for HIV". The items were scored on a 5-point scale ranging from - 2 (strongly disagree) to +2 (strongly agree) with positive values indicating healthier intentions. Participants had the option to respond "not sure" which was given a neutral score of 0. Higher scores equal greater intentions to get tested for HIV. The total range for scores was -14 to 14.
Time Frame: Baseline, 4 weeks, 3 months and 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
score on a scale
  Baseline | 0.14 (0.83) | 0.06 (0.82)
  4 Weeks | 0.57 (0.87) | 0.05 (0.85)
  3 Months | 0.55 (0.81) | 0.07 (0.85)
  6 Months | 0.55 (0.93) | 0.11 (0.88)

3. Secondary Outcome: Number of Students Tested for HIV at Month 1
Description: The number of participants tested for HIV was measured by tracking data reported by school-based health center staff. The school-based health center staff recorded (by study Id number) if participant came in for testing in the last month and the date of the test.
Time Frame: Month 1
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 1 | 0

4. Secondary Outcome: Number of Students Tested for HIV at Month 2
Description: as for outcome 3
Time Frame: Month 2
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 1 | 0

5. Secondary Outcome: Number of Students Tested for HIV at Month 3
Description: as for outcome 3
Time Frame: Month 3
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 0 | 0

6. Secondary Outcome: Number of Students Tested for HIV at Month 4
Description: as for outcome 3
Time Frame: month 4
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 0 | 0

7. Secondary Outcome: Number of Students Tested for HIV at Month 5
Description: as for outcome 3
Time Frame: Month 5
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 0 | 0

8. Secondary Outcome: Number of Students Tested for HIV at Month 6
Description: as for outcome 3
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
Participants | 1 | 0

9. Secondary Outcome: Knowledge About HTC
Description: Participants' knowledge about HTC was measured with 12 questions (e.g., "If you are tested for HIV, you have to wait a long time to find out the results" and "The earlier HIV is caught, the better chance a person has of effectively managing the virus"). Participants responded true, false, or not sure. Responses were recoded into 1 (correct) or 0 (incorrect; responses of "not sure" were coded as incorrect) and a sum of all 12 items was calculated to provide a HTC knowledge score for each participant (Total range was from 0 to 12.) Higher values represent higher knowledge around HTC.
Time Frame: Baseline, 4 weeks, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
score on a scale
  Baseline | 8.18 (2.68) | 7.74 (3.11)
  4 Weeks | 10.01 (3.09) | 8.15 (3.32)
  3 Months | 9.91 (3.06) | 7.92 (3.61)
  6 Months | 9.93 (3.25) | 8.26 (3.54)

10. Secondary Outcome: Self-efficacy Around HIV Testing and Counseling
Description: Self-efficacy for HTC was assessed with 4 items, rated on a confidence scale (e.g., "How confident are you that you could find information about how and where you can get STI and/or HIV testing?"). The total range was from 0-100. A higher score indicates a higher level of self-efficacy around HTC. A mean of the 4 items was calculated for each participant with higher scores indicating higher self-efficacy for HTC.
Time Frame: Baseline, 4 weeks, 3 months, 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
score on a scale
  Baseline | 60.49 (24.87) | 57.80 (24.38)
  4 Weeks | 70.91 (24.80) | 59.24 (25.87)
  3 Months | 69.84 (23.46) | 58.11 (27.95)
  6 Months | 69.93 (26.54) | 58.93 (29.34)

11. Secondary Outcome: Self-efficacy Around Overall Health
Description: Self-efficacy for managing overall health was assessed with 4 items, rated on a 100% confidence scale (e.g., "How confident are you that you could discuss your health concerns with a health provider?"). The total range was from 0-100%.A mean of the 4 items was calculated for each participant with higher scores indicating higher self-efficacy for managing overall health.
Time Frame: Baseline, 4 weeks, 3 months, 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlayTest! Game | Control Games
Number analyzed (Participants) | 145 | 142
score on a scale
  Baseline | 76.84 (22.47) | 73.33 (25.59)
  4 Weeks | 78.00 (24.12) | 71.09 (26.45)
  3 Months | 75.53 (25.29) | 68.31 (29.21)
  6 Months | 76.53 (24.45) | 69.36 (29.77)

12. Secondary Outcome: HIV Testing and Counseling Behavior (Self-Report)
Description: At each time point the participants indicated whether they had ever been tested for HIV with the response options: yes, no, not sure, and decline to answer.
Time Frame: Baseline, 4 Weeks, 3 Months, 6 Months
Population: The number of overall analyzed at the different timepoints after baseline differ from the baseline numbers due to the fact that some participants missed the assessment time point window and did not complete the assessment; therefore those data points are missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  Baseline: Yes | 12 | 9
  Baseline: No | 108 | 113
  Baseline: Decline to Answer | 5 | 3
  Baseline: Not sure | 20 | 17
  4 Weeks: number analyzed (Participants) | 143 | 135
  4 Weeks: Yes | 12 | 8
  4 Weeks: No | 106 | 107
  4 Weeks: Decline to Answer | 5 | 3
  4 Weeks: Not sure | 20 | 17
  3 Months: number analyzed (Participants) | 137 | 128
  3 Months: Yes | 10 | 7
  3 Months: No | 103 | 101
  3 Months: Decline to Answer | 5 | 3
  3 Months: Not sure | 19 | 17
  6 Months: number analyzed (Participants) | 139 | 129
  6 Months: Yes | 11 | 7
  6 Months: No | 104 | 103
  6 Months: Decline to Answer | 5 | 3
  6 Months: Not sure | 19 | 16

13. Secondary Outcome: Perceived Barriers to HIV Testing
Description: Perceived Barriers was measured with a one question instrument that asks participants what reasons would most likely keep them from getting tested if they thought they had HIV (examples of options were "I don't know where to go", "It costs too much"). The instrument allowed participants to select all reasons that apply.
Time Frame: Baseline
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 57 | 67
  Outpatient clinic too far away | 15 | 13
  Costs too much | 39 | 39
  No time to get tested | 15 | 22
  Test pain/uncomfortable | 57 | 54
  Embarrasment | 88 | 82
  Someone might recognize me | 60 | 63
  Parents would find out | 92 | 89
  Boyfriend/girlfriend might find out | 35 | 39
  Parents' permission (afraid to ask) | 52 | 48
  Don't want to know if I have HIV | 30 | 26
  Friends might find out | 30 | 26
  Too much trouble | 11 | 16
  Little I can do if I have HIV | 31 | 29
  Other | 10 | 10

14. Secondary Outcome: Perceived Barriers to HIV Testing
Description: as for outcome 13
Time Frame: 4 weeks
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 23 | 53
  Outpatient clinic too far away | 9 | 16
  Costs too much | 17 | 41
  No time to get tested | 21 | 24
  Test pain/uncomfortable | 16 | 47
  Embarrasment | 81 | 82
  Someone might recognize me | 52 | 58
  Parents would find out | 67 | 79
  Boyfriend/girlfriend might find out | 24 | 29
  Parents' permission (afraid to ask) | 35 | 46
  Don't want to know if I have HIV | 21 | 20
  Friends might find out | 21 | 20
  Too much trouble | 7 | 13
  Little I can do if I have HIV | 18 | 21
  Other | 7 | 4

15. Secondary Outcome: Perceived Barriers to HIV Testing
Description: as for outcome 13
Time Frame: 3 months
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 27 | 50
  Outpatient clinic too far away | 12 | 14
  Costs too much | 22 | 43
  No time to get tested | 18 | 29
  Test pain/uncomfortable | 13 | 45
  Embarrasment | 77 | 74
  Someone might recognize me | 51 | 62
  Parents would find out | 65 | 71
  Boyfriend/girlfriend might find out | 23 | 29
  Parents' permission (afraid to ask) | 31 | 44
  Don't want to know if I have HIV | 18 | 20
  Friends might find out | 18 | 20
  Too much trouble | 11 | 14
  Little I can do if I have HIV | 23 | 15
  Other | 6 | 8

16. Secondary Outcome: Perceived Barriers to HIV Testing
Description: as for outcome 13
Time Frame: 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 28 | 47
  Outpatient clinic too far away | 12 | 20
  Costs too much | 19 | 42
  No time to get tested | 31 | 25
  Test pain/uncomfortable | 22 | 43
  Embarrasment | 81 | 69
  Someone might recognize me | 55 | 59
  Parents would find out | 74 | 69
  Boyfriend/girlfriend might find out | 26 | 33
  Parents' permission (afraid to ask) | 40 | 45
  Don't want to know if I have HIV | 20 | 19
  Friends might find out | 20 | 19
  Too much trouble | 11 | 11
  Little I can do if I have HIV | 21 | 25
  Other | 5 | 6

17. Secondary Outcome: Perceived Barriers to STI Testing
Description: Perceived Barriers was measured with a one question instrument that asks participants what reasons would most likely keep them from getting tested if they thought they had an STI (examples of options were "I don't know where to go", "It costs too much"). The instrument allowed participants to select all reasons that apply.
Time Frame: Baseline
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 58 | 62
  Outpatient clinic too far away | 13 | 17
  Costs too much | 42 | 46
  No time to get tested | 12 | 22
  Test pain/uncomfortable | 50 | 51
  Embarrasment | 85 | 90
  Someone might recognize me | 56 | 63
  Parents would find out | 87 | 92
  Boyfriend/girlfriend might find out | 31 | 34
  Parents' permission (afraid to ask) | 65 | 60
  Don't want to know if have STI | 33 | 26
  Friends might find out | 58 | 46
  Too much trouble | 12 | 18
  Little I can do if I have a STI | 31 | 26
  Other | 11 | 11

18. Secondary Outcome: Perceived Barriers to STI Testing
Description: as for outcome 17
Time Frame: 4 weeks
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 26 | 53
  Outpatient clinic too far away | 11 | 13
  Costs too much | 21 | 42
  No time to get tested | 25 | 21
  Test pain/uncomfortable | 18 | 46
  Embarrasment | 78 | 81
  Someone might recognize me | 52 | 58
  Parents would find out | 71 | 75
  Boyfriend/girlfriend might find out | 26 | 32
  Parents' permission (afraid to ask) | 41 | 53
  Don't want to know if have STI | 23 | 20
  Friends might find out | 38 | 47
  Too much trouble | 13 | 12
  Little I can do if I have a STI | 13 | 22
  Other | 8 | 4

19. Secondary Outcome: Perceived Barriers to STI Testing
Description: as for outcome 17
Time Frame: 3 months
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 30 | 40
  Outpatient clinic too far away | 11 | 14
  Costs too much | 19 | 42
  No time to get tested | 28 | 29
  Test pain/uncomfortable | 13 | 38
  Embarrasment | 71 | 74
  Someone might recognize me | 50 | 60
  Parents would find out | 63 | 72
  Boyfriend/girlfriend might find out | 20 | 26
  Parents' permission (afraid to ask) | 33 | 49
  Don't want to know if have STI | 14 | 23
  Friends might find out | 35 | 40
  Too much trouble | 11 | 15
  Little I can do if I have a STI | 20 | 17
  Other | 4 | 8

20. Secondary Outcome: Perceived Barriers to STI Testing
Description: as for outcome 17
Time Frame: 6 months
Population: Only participants that completed the study were analyzed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Active Game | Control Game
Number analyzed (Participants) | 145 | 142
Participants
  I don't know where to go | 28 | 48
  Outpatient clinic too far away | 17 | 20
  Costs too much | 23 | 46
  No time to get tested | 36 | 30
  Test pain/uncomfortable | 19 | 41
  Embarrasment | 75 | 72
  Someone might recognize me | 58 | 59
  Parents would find out | 76 | 72
  Boyfriend/girlfriend might find out | 23 | 31
  Parents' permission (afraid to ask) | 46 | 48
  Don't want to know if have STI | 19 | 17
  Friends might find out | 36 | 37
  Too much trouble | 11 | 16
  Little I can do if I have a STI | 21 | 19
  Other | 5 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 6 months.
Arm/Group | PlayTest! Game | Control Games
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/142
Other Adverse Events (participants affected / at risk) | 0/145 | 0/142

LIMITATIONS AND CAVEATS:
This study was impacted by COVID. Please refer to attached data analysis document that highlights how COVID impacted the project and data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03713034/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT03713034/ICF_001.pdf